CLINICAL TRIAL: NCT00681200
Title: Mechanisms of Meditation in Hypertension in Blacks
Brief Title: Evaluating Mechanisms of Blood Pressure Reduction Using Meditation in Hypertensive African Americans
Acronym: HMEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Howard University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director, Center for Natural Medicine and Prevention, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 602; R01HL083944-01A1 (NIH); NCT00681200 (Registry Identifier: Clinical Trials.gov)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
Keywords: Blood Pressure Reduction; Stress Reactivity and Recovery; Meditation; Transcendental Meditation; Stress Reduction; Stress Management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced health education program (Active Comparator): This active treatment group consists of classes in health education and a social support group to enhance participant motivation and positive reinforcement to make healthier lifestyle choices (e.g. wholesome diet, increased exercise, reduced salt intake, and decreased use of alcohol and smoking). Note that this comparison group does not have a stress management component.
  Interventions: Behavioral: Enhanced health education
- Transcendental Meditation program (Experimental): Transcendental Meditation program plus health education. Basic American Heart Association (AHA) recommendations for lifestyle modification to reduce risk of heart disease will be given in a didactic classroom context.
  Interventions: Behavioral: Transcendental Meditation program

INTERVENTIONS:
Behavioral: Enhanced health education — health education and social support
  Arms: Enhanced health education program
Behavioral: Transcendental Meditation program — The TM program plus didactic-based health education classes
  Arms: Transcendental Meditation program

SUMMARY:
High blood pressure is a common health problem among people in the United States. This study will compare the effectiveness of a meditation program versus a health education program at decreasing stress and lowering blood pressure levels among African-American adults with high blood pressure.

DETAILED DESCRIPTION:
Hypertension, also known as high blood pressure, is one of the most common health problems among adults, particularly African Americans. If left untreated, it can lead to heart failure, kidney failure, or stroke. High blood pressure can be caused by many factors, including stress, diet, diabetes, kidney disease, or obesity. Typical treatments include taking medication, losing weight, and quitting smoking. Meditation may also be an effective way to decrease stress levels and lower blood pressure. This study will examine the effects of a specific type of meditation, Transcendental Meditation (TM), on stress and blood pressure levels. In previous studies, TM has been shown to have a positive effect on reducing blood pressure levels, but more research is needed to confirm these benefits. This study will compare the effectiveness of a TM program with an enhanced health education (EHE) program for reducing stress and blood pressure levels in African Americans with high blood pressure.

This 4-month study will enroll African Americans with early stage hypertension. Recruiting will be conducted from Howard University Medical Center in Washington, DC. First, participants will take part in 3 days of baseline testing, including a medical history review, blood pressure and heart rate measurements, an echocardiogram to obtain images of the heart, and blood and urine collection. Over a 24-hour period, blood pressure and heart rate will be measured continuously and participants will wear a pedometer to keep track of the distance they walk. Participants will also complete a stress test; a treadmill exercise test; and questionnaires on mental health, physical health, and lifestyle.

After the 3-day baseline period, participants will attend an informational meeting with the study staff and other study participants. They will then be randomly assigned to either the TM group or the EHE group. Participants in the TM group will learn a simple meditation technique over a 6-day period. They will be expected to meditate for 20 minutes twice a day for 4 months. Participants will attend follow-up meetings with a meditation instructor every 2 weeks throughout the study, and they will record their progress in a daily diary. Participants in the EHE program will take part in 14 events during the study, including watching educational films, listening to guest speakers, and participating in other instructional activities that will provide health information about blood pressure regulation. In addition, all participants will attend standard health education classes every 2 weeks. These classes will provide information about reducing the risk factors related to heart disease and stroke. Once a month, participants will attend a study visit and undergo blood pressure and heart rate measurements. At the end of the 4-month study period, all participants will undergo repeat baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as African American
* Resides in Washington, DC or surrounding communities
* Has stage I hypertension, defined as systolic blood pressure between 140 and 159 mm Hg and/or diastolic blood pressure between 90 and 99 mm Hg, on average, without taking antihypertensive medications in the sympatholytic class (e.g., beta blockers, alpha antagonists, central nervous system agonists)

Exclusion Criteria:

* Blood pressure levels of less than 140/90 mm Hg or greater than 160/100 mm Hg
* History of clinical cardiovascular disease (e.g., heart attack, angina, intermittent claudication, congestive heart failure, stroke)
* Long-term kidney failure
* Any other life-threatening illness (e.g., advanced cancer)
* History of major psychiatric disorder (e.g., psychosis, dementia, substance abuse disorder)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
In-clinic and ambulatory blood pressure | Measured at Month 4

SECONDARY OUTCOMES:
Cardiovascular hemodynamics and stress hormones | Measured at Month 4
telomerase gene expression | 4 months
  telomerase gene expression as measured HTERT and HTR

CONTACTS AND LOCATIONS:
Overall Officials: Otelio Randall, MD, Principal Investigator — Howard University
Locations (1):
- Howard University College of Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
outside investigators may contact the study PIs for sharing of the database

REFERENCES:
- [Result] Duraimani SLC (2012) Lifestyle Modifications and Healthy Biological Aging: Effects of Telomerase Activity and Telomere Length. Ann Arbor Mich: Dissertation Information Service
- [Result] Duraimani S, Schneider RH, Randall OS, Nidich SI, Xu S, Ketete M, Rainforth MA, Gaylord-King C, Salerno JW, Fagan J. Effects of Lifestyle Modification on Telomerase Gene Expression in Hypertensive Patients: A Pilot Trial of Stress Reduction and Health Education Programs in African Americans. PLoS One. 2015 Nov 16;10(11):e0142689. doi: 10.1371/journal.pone.0142689. eCollection 2015. PMID 26571023